CLINICAL TRIAL: NCT04619472
Title: A Multicenter, Single Group Target Value Clinical Study to Evaluate Safety and Effectiveness of Radiofrequency Ablation System in the Treatment of Peripheral Lung Tumors
Brief Title: Safety and Effectiveness of Radiofrequency Ablation System in the Treatment of Peripheral Lung Tumors
Acronym: BRONC-RFⅡ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Broncus Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-RF-01
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-04

CONDITIONS: Lung Neoplasms; Pulmonary Metastasis
Keywords: Lung Neoplasms; Radiofrequency ablation; Pulmonary Metastasis; Primary Pulmonary Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency Ablation (RFA) (Experimental): The subjects will first undergo interventional bronchoscopy to reach the target lesion through the bronchial pathway. Then the lung lesions will be treated with radiofrequency ablation using the pulmonary radiofrequency ablation system and the disposable pulmonary radiofrequency ablation catheter.
  Interventions: Device: Pulmonary Radiofrequency Ablation System and the Disposable Pulmonary Radiofrequency Ablation Catheter

INTERVENTIONS:
Device: Pulmonary Radiofrequency Ablation System and the Disposable Pulmonary Radiofrequency Ablation Catheter — The conjunction of the pulmonary RFA system with the disposable pulmonary RFA catheter developed by Hangzhou Broncus Medical Co., Ltd. is aim to specifically target lung tumors. The ablation catheter is designed to reach the tumor through the bronchial pathway.

SUMMARY:
It is a multicenter, single group target value clinical trial to evaluate the safety and effectiveness of radiofrequency ablation for peripheral lung tumors under the conjunction of the pulmonary radiofrequency ablation system with the disposable pulmonary radiofrequency ablation catheter developed by Hangzhou Broncus Medical Co., Ltd.

DETAILED DESCRIPTION:
The subjects will first undergo interventional bronchoscopy to reach the target lesion through the bronchial pathway. Then the lung lesions will be treated with radiofrequency ablation using the pulmonary radiofrequency ablation system and the disposable pulmonary radiofrequency ablation catheter. During the study, eligible subjects will be followed up intraoperatively, 24 hours after operation, before discharge/ 7 days after operation (whichever occurs first), 30 days (±7 days) after operation, 3 months (±7 days) after operation, 6 months (±15 days) after operation, 9 months (±15 days) after operation, and 12 months (±15 days) after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Planned ablated main lesions are pathologically confirmed and other planned ablated lesions are pathologically confirmed or clinical evaluated as primary NSCLC or pulmonary metastasis, and the primary lesions of lung metastasis subjects has been well controlled;
3. Number of unilateral lung lesions: ≤ 3 (excepting for multiple primary lung cancers);
4. Each lung lesion in size: ≤3 cm ;
5. Subjects refuse surgery or are considered intolerant of surgery;
6. Subjects refuse or are considered unsuitable for radiotherapy/chemotherapy, or are non-responders for previous radiotherapy/chemotherapy, or has disease progression after radiotherapy/chemotherapy;
7. It is feasible to arrive at the target lesions through bronchus path and carry out ablation operations, assessed by investigators;
8. Subjects whose Eastern oncology cooperative group (ECOG) physical state score: ≤3;
9. Subjects agree to undergo radiofrequency ablation to treat pulmonary lesions.

Exclusion Criteria:

1. Subjects with severe bleeding tendency and irreversible clotting disorders; or subjects who have stopped anticoagulation therapy and/or antiplatelet drugs for less than 7 days before ablation;
2. Subjects whose preoperative examination within 1 month shows intrathoracic lymph node or extra-pulmonary metastasis (except for extra-pulmonary metastasis controlled by local therapy);
3. Planned ablated lesions have received radiotherapy within past 6 months;
4. Subjects with high-risk disease for ablation operation;
5. The nearest distance between the tumors and trachea, main bronchial tube, esophagus, aortic arch branch, main pulmonary artery, left and right pulmonary artery and the heart is less than 2cm;
6. Subjects who have participated in the last 30 days or is participating in other clinical studies;
7. Subjects who are pregnant or have pregnancy plan during the study;
8. Subjects with bronchoscopy contraindications;
9. Subjects with implantable cardiac pacemakers, implantable defibrillators, or other active implants;
10. Subjects with general anesthesia contraindications;
11. Subjects with other conditions that need to be excluded as determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Complete ablation rate of main lesions at 6 months | Six months
  Six months after the overall ablation procedure, the proportion that subjects whose main lesions maintain completely ablated account for all evaluable subjects who receive radiofrequency ablation.

SECONDARY OUTCOMES:
Technical success rate (in terms of ablation operations) | Immediately after Each Operation
  It is defined as the proportion that the ablation operations in which the test device is successfully placed at the target lesion and the device is successfully withdrawn after treatment procedure, account for all ablation operations.
Complete ablation rate at 6 months (in terms of ablation lesions) | Six months
  Six months after overall ablation procedure, the proportion that lesions completely ablated account for all evaluable lesions that receive radiofrequency ablation.
Complete ablation rate at 6 months (in terms of subjects) | Six months
  Six months after overall ablation procedure, the proportion that subjects whose all ablation lesions maintain completely ablated account for all evaluable subjects who receive radiofrequency ablation.
Intrapulmonary progression-free survival rate at 6 months | Six months
  Six months after overall ablation procedure, the proportion that subjects with no progression in the lung (the original ablation lesions maintain completely ablated, no metastasis of hilar lymph nodes, and no new lesions) account for all evaluable subjects who receive radiofrequency ablation.
Complete ablation rate at 12 months (in terms of ablation lesions) | Twelve months
  Twelve months after the completion of the overall ablation, the proportion that lesions which maintain completely ablated account for all evaluable lesions that receive radiofrequency ablation.
Complete ablation rate at 12 months (in terms of subjects) | Twelve months
  Twelve months after overall ablation procedure, the proportion that subjects whose all ablation lesions maintain completely ablated account for all evaluable subjects who receive radiofrequency ablation.
Intrapulmonary progression-free survival rate at 1 year | Twelve months
  Twelve months after the completion of the overall ablation, the proportion that subjects with no progression in the lung (the original ablation lesions maintain completely ablated, no metastasis of hilar lymph nodes, and no new lesions) account for all evaluable subjects who receive radiofrequency ablation.
Overall survival rate (OS) at 1 year | Twelve months
  It is defined as the proportion of surviving subjects at 1 year from enrollment.
Quality of life (QoL) | Twelve months
  The QoL changes are evaluated according to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORCT QLQ C30) assessment scale during the follow-up. The EORCT QLQ C30 incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease.
Safety | Twelve months
  All adverse events will be recorded during operation and during the follow-up, and be evaluated according to the CTCAE v5.0 (if applicable). Related and possible related AEs and SAEs will be determined and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (3):
- China (3):
  - The First Hospital of Peking University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No